CLINICAL TRIAL: NCT02977234
Title: Hysteroscopic Tubal Occlusion With the Use of Iso Amyl-2-cyanoacrylate in Patients With Hydrosalpinx
Brief Title: Hysteroscopic Tubal Occlusion Using Iso-Amyl 2-Cyano Acrylate (Amcrylate) in Patients With Hydrosalpinx
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed I Amer, Professor, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ASU123
Record Dates: First submitted 2016-11-23; First posted 2016-11-30 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Hydrosalpinx; Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — isoamyl 2-cyanoacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iso-Amyl 2-Cyano Acrylate (Experimental): Hysteroscopic Tubal Occlusion Using Iso-Amyl 2-Cyano Acrylate (Amcrylate) in Patients With Hydrosalpinx
  Interventions: Drug: Isoamyl 2-Cyanoacrylate

INTERVENTIONS:
Drug: Isoamyl 2-Cyanoacrylate

SUMMARY:
The purpose of this study is to assess the effectiveness of hysteroscopic tubal application of Iso Amyl-2-cyanoacrylate in occluding uterine tubes of infertile women with hydrosalpinx, which would make it an easy approach for occluding tubes with hydrosalpinx prior to IVF.

DETAILED DESCRIPTION:
The study will be conducted according to the guidelines on human experimentation of the 1975 Declaration of Helsinki. For all patients after taking signed informed consent , transcervical hysteroscopic cannulation of the proximal one centimeter of fallopian tubes with hydrosalpinx, will be done using a 4 Fr, 42cm long, polyethylene ureteric catheter, where 0.5 ml of Iso Amyl-2-cyanoacrylate (AMCRYLATE®) will be injected.

All the surgical procedures will be performed without anesthesia, only premedication with an NSAID (e.g. NaproxenR) is given orally one hour before the procedure.

Each patient will be under close observation for the first 24 hours postprocedure for any signs of inflammation as abdominal pain, tenderness or fever and for the vital data.

Hysterosalpingography will be done for all patients 0ne and 3 months postinjection to confirm tubal occlusion prior to IVF.

ELIGIBILITY:
Inclusion Criteria:

Infertile women due to tubal factor with hydrosalpinx (unilateral or bilateral) prepared for IVF.

Exclusion Criteria:

1. Acute Pelvic inflammatory disease.
2. Intra uterine pathology

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Fallopian tubal occlusion in patients with hydrosalpinx. | from one to three months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Amer, MD, Principal Investigator — Ain Shams University maternity hospital
Locations (1):
- AIn Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided